CLINICAL TRIAL: NCT04709367
Title: Characterization of Residual Limb Volume Changes in Transfemoral Amputees: Descriptive Prospective Longitudinal Observational Study.
Brief Title: Characterization of Residual Limb Volume Changes in Transfemoral Amputees
Status: Completed | Type: Observational
Sponsor: Istituto Nazionale Assicurazione contro gli Infortuni sul Lavoro (Other)
Collaborators: Scuola Superiore Sant'Anna di Pisa (Other)
Responsible Party: Sponsor
Other Study IDs: P-PPRAI1/2-01
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2021-01-14 (Actual); Status verified 2021-01

CONDITIONS: Amputation Stump
Keywords: Amputee; Prosthetic socket; Transfemoral residual limb; Volume change; 3D scan

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: 3D optical scan — The clinical protocol consisted of four test sessions in four different days for an overall duration of 3 weeks. During the 1st session, amputees' residual limb volume was measured 7 times at intervals of 10 minutes after the prosthesis removal. During the subsequent sessions, the residual limb volume was measured immediately after the prosthesis doffing and after the amputee's stabilization time, before and after 15-min of walking on a treadmill, both in the morning and in the afternoon.

SUMMARY:
This study quantifies residual limb volume fluctuations affecting transfemoral amputees due to the prosthesis doffing, physical activity, and testing time.

DETAILED DESCRIPTION:
The first test session aims at measuring residual limb volume at 7 time-points, with 10 minute intervals, after prosthesis doffing. This allows for evaluating the time required for volume stabilization after prosthesis removal, for each amputee. In subsequent sessions, 16 residual limb scans in a day for each amputee are captured to evaluate volume changes due to prosthesis removal and physical activity, in two times per day (one in the morning, one in the afternoon). These measurements are repeated in three different days, a week apart from each other, for a total of 48 scans for each amputee.

ELIGIBILITY:
Inclusion Criteria:

* Stabilized (i.e., time since amputation > 18 months) transfemoral amputees
* Age between 18 and 65 years old
* Subjects able to safely perform the physical tasks required in the experimental protocol
* Subjects provided with prostheses

Exclusion Criteria:

* Denial of informed consent to participate in the study
* Inability to maintain the required position during the 3D scanning for at least 5 minutes
* Concomitant general or localized comorbidities / disabilities, which may interfere with the study
* Pathological conditions affecting the residual limb
* Allergy / sensitivity with polydimethylsiloxane (PDMS)
* Pathological cardiopulmonary / cardiovascular conditions
* Pregnancy or breastfeeding
* Presence of psychiatric co-morbidities
* Presence of cognitive deficits which may compromise the understanding of the required tasks
* Difficulty in understanding the Italian language
* Insufficient degree of collaboration
* Consumption of alcohol or diuretics before tests

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: transfemoral amputees
Sampling Method: Non-Probability Sample
Enrollment: 24 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2020-08-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
Residual limb volume changes | The protocol consisted of four test sessions in four different days for an overall duration of 3 weeks
  Residual limb volume changes due to prosthesis doffing, physical activity, and testing time are measured by a proper experimental set-up, including a 3D metrology-grade optical scanner.

SECONDARY OUTCOMES:
Pressure distribution at the prosthetic socket - residual limb interface | The protocol consisted of four test sessions in four different days for an overall duration of 3 weeks
  Pressure distributions at the residual limb/ socket interface are measured by the F-Socket Pressure Measurement System, during:
  * Walking (five gait cycles, three times);
  * Walking up and down slope (five gait cycles, three times);
  * Walking upstairs and downstairs (six stairs cycles, three times);
  * Sitting down and up (three times).

CONTACTS AND LOCATIONS:
Overall Officials: Emanuele Gruppioni, Principal Investigator — INAIL Prosthesis Centre
Locations (1):
- INAIL Prosthesis Centre, Bologna, BO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Paterno L, Truppa L, Ibrahimi M, Rosini E, Gruppioni E, Ricotti L, Menciassi A. Quantitative analysis of interface pressures in transfemoral prosthetic sockets. Prosthet Orthot Int. 2024 Apr 1;48(2):176-183. doi: 10.1097/PXR.0000000000000251. Epub 2023 Jun 28. PMID 37379468
- [Derived] Paterno L, Ibrahimi M, Rosini E, Menfi G, Monaco V, Gruppioni E, Ricotti L, Menciassi A. Residual limb volume fluctuations in transfemoral amputees. Sci Rep. 2021 Jun 10;11(1):12273. doi: 10.1038/s41598-021-91647-9. PMID 34112873